CLINICAL TRIAL: NCT03737604
Title: Transversus Abdominis Plane (TAP) Blocks With Ropivacaine Continuous Infusion Catheters vs Single Dose Liposomal Bupivicaine: A Prospective Randomized Control Trial for Pain Control After Renal Transplant Surgery
Brief Title: TAP Blocks With Ropivacaine Continuous Infusion Catheters vs Single Dose Liposomal Bupivicaine After Kidney Transplant
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205738
Record Dates: First submitted 2018-10-09; First posted 2018-11-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Transplant;Failure,Kidney; Pain, Postoperative
Keywords: Transversus Abdominis Plane Block; Ropivacaine; Liposomal bupivacaine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Masking Description: Unable to mask based on physical characteristics of liposomal bupivacaine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine Continuous Infusion Catheter (Active Comparator): Ropivacaine Continuous Infusion Catheter: ultrasound guided TAP block and TAP catheter placement performed with 0.2% ropivacaine (2.5 mg/kg) and maintained with 0.2% ropivacaine infusion 8 ml/hour via catheter.
  Interventions: Drug: Ropivacaine Continuous Infusion Catheter
- Single dose liposomal bupivicaine (Active Comparator): Liposomal bupivacaine TAP block: ultrasound guided TAP block a performed with up to 12 ml 0.25% bupivacaine and prolonged with liposomal bupivacaine 133 mg diluted to total volume of 20 ml with preservative free saline.
  Interventions: Drug: Single Dose Liposomal Bupivicaine

INTERVENTIONS:
Drug: Ropivacaine Continuous Infusion Catheter — For those randomized to the TAP catheter group, ultrasound guidance will be used for TAP block and 5mls 1% lidocaine will be used for skin infiltration. A peripheral nerve catheter will be placed approximately 3-5 cm into the TAP space after injection of the ropivacaine solution. A bolus dose of 2.5 mg/kg of ropivacaine will be administered in a volume of 30 ml up to a maximum of 150 mg. An infusion with a programmable pump will be initiated at a rate of 8 ml/hr of 0.2% ropivacaine on the inpatient floor.
  Other Names: TAP block initiated with ropivacaine bolus and infusion
  Arms: Ropivacaine Continuous Infusion Catheter
Drug: Single Dose Liposomal Bupivicaine — TAP block will be performed using ultrasound guidance. 12ml of 0,25% plain bupivacaine will be used for skin infiltration and to open up the TAP. Liposomal bupivacaine 266 mg (1.3% in 20 ml) will be diluted to 40 ml volume with 20 ml of preservative free normal saline. 20 ml (133mg) of liposomal bupivicaine will then be injected into the TAP.
  Other Names: TAP block with liposomal bupivacaine
  Arms: Single dose liposomal bupivicaine

SUMMARY:
This study is a comparison of the analgesic efficacy of transversus abdominis plane (TAP) blocks with ropivacaine bolus plus continuous ropivacaine infusion via catheters versus single shot TAP blocks with liposomal bupivacaine.

DETAILED DESCRIPTION:
This study is a comparison of the analgesic efficacy of TAP blocks provided by ropivacaine bolus plus continuous ropivacaine infusion via catheters versus single shot TAP blocks with liposomal bupivacaine.

In the Liposomal Bupivacaine group, TAP block will be performed using ultrasound guidance. 12ml of 0,25% plain bupivacaine will be used for skin infiltration and to open up the TAP. Liposomal Bupivacaine 266 mg (1.3% in 20 ml) will be diluted to 40 ml volume with 20 ml of preservative free normal saline. 20 ml (133mg) of liposomal bupivicaine will then be injected into the TAP.

For those randomized to the TAP catheter group, ultrasound guidance will be used for TAP block and 5 mls 1% lidocaine will be used for skin infiltration. A peripheral nerve catheter will be placed approximately 3-5 cm into the TAP space after injection of ropivacaine. A bolus dose of 2.5 mg/kg of ropivacaine will be administered in a volume of 30 ml up to a maximum of 150 mg. An infusion with a programmable pump will be initiated at a rate of 8 ml/hr of 0.2% ropivacaine on the inpatient floor.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 years or older
* Renal Transplant Recipients

Exclusion Criteria:

* Patients less than 18 years of age
* Pregnant Women
* Prisoners
* Opioid Tolerant Patients taking more than 30 mg/day of oral morphine equivalent analgesia
* Patients on Systemic anti coagulation
* Patients unable to provide consent
* Hypersensitivity to amide-type local anesthetic or any component of the drug formula

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Total Opioid Consumption | Through 4 days following renal transplant surgery
  Total amount of opioid analgesic administered following renal transplant surgery converted using standard equivalency calculations to morphine equivalents mg/kg

SECONDARY OUTCOMES:
Proportion of pain scores indicating severe pain | Through 4 days following renal transplant surgery
  Proportion of pain scores 7 or higher indicating severe pain as determined by patient report of pain using verbal pain score from 0 (no pain) to10 (most severe pain)
Post Operative Nausea | Through 4 days following renal transplant surgery
  Count of post operative nausea episodes
Post Operative Vomiting | Through 4 days following renal transplant
  Count of post operative vomiting events
Respiratory Depression | Through 4 days following renal transplant surgery
  Count of Respiratory Depression events defined as respiratory rate less than 8 breaths per minute
Post Operative Care Unit and Hospital Length of Stay | Up to 2 weeks following renal transplant surgery
  Length of Stay
Acquisition Costs Related to Analgesia | Up to 2 weeks following renal transplant surgery
  Analgesia Related Costs defined as the sum of hospital specific costs to acquire medications and supplies needed to perform block or administer analgesic and local anesthetic medications

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-experimental-medicine-ropivacaine-for-pain-control-after-kidney-transplant-995191/